CLINICAL TRIAL: NCT00260104
Title: Risk Factors of Individuals With Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Other Study IDs: ICP058
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2008-05-26 (Estimated); Status verified 2008-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
It would be useful to study coronary arteriovenous difference of various markers in patients who are undergoing coronary angiography for suspected coronary artery disease. Environmental and genetic factors may play a role in the progression of coronary artery disease. The goal of this project is to establish a series of cross-sectional / case-control studies to evaluate risk factors of coronary artery disease in China.

DETAILED DESCRIPTION:
This study is designed to investigate the epidemiologic, genetic, laboratory and clinical characterization of individuals with coronary artery disease. The study group will consist of consecutive patients who are undergoing coronary angiography for suspected coronary artery disease. The diagnosis of coronary artery disease will be confirmed by coronary angiography performed with the Judkins technique using a quantitative coronary angiographic system. Coronary artery disease will be considered to be present if there is a diameter stenosis of at least 50% in at least one of the three major epicardial coronary arteries. The number of diseased vessels will be determined and a classification of 1-, 2-, and 3-vessel disease will be used. Coronary artery segments will be defined according to the Coronary Artery Surgery Study classification. Blood samples from vein and coronary artery will be collected. We will study coronary arteriovenous difference of various markers. Urinary samples will be obtained the day of coronary angiography. We will explore the environmental (including family history, life style, diet, physical activity, neuropsychological functioning，plasma levels of oxidative stress factors, angiogenic factors, and inflammatory markers, etc.) and genetic (including oxidative stress factors and inflammatory factors, etc.) risk factors. We will study the association between various environmental risk factors with the clinical characterization and correlation between the genetic polymorphisms and the presence of coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* This is a study only of Chinese.
* Subjects will be allowed to participate if they self-identify as Chinese.
* The age range of the participants will be between 18 and 89 years.
* The study group will consist of consecutive patients who are undergoing coronary angiography for suspected coronary artery disease.

Exclusion Criteria:

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Bin Wang, Ph.D, Principal Investigator — Department of Pharmacology, Institute of Clinical Pharmacology, Nanjing Medical University
Locations (1):
- Nanjing Medical University, Nanjing, China

REFERENCES:
- [Result] Tang NP, Wang LS, Yang L, Gu HJ, Zhu HJ, Zhou B, Sun QM, Cong RH, Wang B. Preproghrelin Leu72Met polymorphism in Chinese subjects with coronary artery disease and controls. Clin Chim Acta. 2008 Jan;387(1-2):42-7. doi: 10.1016/j.cca.2007.08.014. Epub 2007 Sep 5. PMID 17884032